CLINICAL TRIAL: NCT02310711
Title: A Pilot Study for the Identification of Targets for Clinical Improvement in Breast Conserving Therapy
Brief Title: Multi-scale Modeling of Breast Conserving Therapy
Acronym: BCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Barbara Bass, Chair, Department of Surgery, The Methodist Hospital Research Institute
Other Study IDs: Pro00006887; IRB0112-0007 (Other: TMHRI IRB); BCTMM01 (Other: Other Protocol ID)
Record Dates: First submitted 2014-12-01; First posted 2014-12-08 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer
Keywords: Breast; Mastectomy; Lumpectomy; Breast Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Standard of Care — Standard of care for early stage breast cancer is breast conserving therapy at this center.
  Other concomitant standard of care treatment • Radiation therapy to the whole breast
  o 45-50 Gy delivered over 25-28 fractions with a boost to the tumor bed of 10-16 Gy delivered over 5-8 fractions

SUMMARY:
The proposed study is a single-center, prospective, pilot, observation study to tabulate and measure the changes that occur during treatment and healing for breast conserving therapy (BCT) in women with non-metastatic breast cancer for comparison to the multiscale model of breast lumpectomy and healing in order to identify targets for improving BCT. The study will be comprised of 12 de novo breast cancer patients with non-metastatic breast cancer undergoing BCT. Subjects will be enrolled in the study during the 3 weeks prior to receiving their BCT surgery and will be followed for six months after the BCT surgery. A total of 6 visits (not including the surgery) are planned.

DETAILED DESCRIPTION:
This is a single-center, prospective, pilot observation study. Eligible subjects who enroll in this study will begin at the time of informed consent, which will occur during the pre-operative, surgical evaluation time. Once consented, a 3-dimensional 180° camera surface image will be taken and a pain-scale score will be completed. Data from the medical history will be recorded. As standard of care, the surgery will be scheduled and performed. Following surgery, a series of 5 standard of care visits will occur over the subsequent 6 months, that will include research measures of local ultrasound x5 and 3-dimensional surface imaging x3. The pain scale score will be administered pre and post ultrasound on the 5 post-operative visits. A judging of the cosmesis will take place at weeks 10 and 26 by independent surgeons. The participant's role in the study will be completed after the week 24 visit.

ELIGIBILITY:
Inclusion Criteria:

1. Adult females ≥ age 30 years
2. Have early stage (Stage I, II), non-metastatic breast cancer
3. Planned to receive BCT
4. Have received a pre-operative mammogram within 30 days of surgery
5. Have received pre-operative magnetic resonance imaging (MRI) within 30 days of surgery
6. Planned to receive post-surgery radiotherapy by whole breast radiotherapy
7. Signed informed consent form prior to any research assessment

Exclusion Criteria:

1. Adult females younger than 30 years of age
2. Previous breast cancer
3. Neo-adjuvant therapy for breast cancer
4. Pregnant or nursing females
5. Participation in a study of investigational drug in the previous 30 days or 5 half-lives of the investigational drug

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer who are having BCT and who satisfy the following criteria will be considered for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2012-05; Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Study Endpoint | Six-month Post-Surgery
  The proportion of subjects with ≥60% agreement between the surgical/healing outcome of the lumpectomy and breast surface contour and the predicted changes from the multi-scale model.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Bass, MD, Principal Investigator — Chair, Department of Sugery
Locations (1):
- Houston Methodist Hopsital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Plan to share data to be determined.

REFERENCES:
- [Background] Salmon R, Garbey M, Moore LW, Bass BL. Interrogating a multifactorial model of breast conserving therapy with clinical data. PLoS One. 2015 Apr 23;10(4):e0125006. doi: 10.1371/journal.pone.0125006. eCollection 2015. PMID 25906048